CLINICAL TRIAL: NCT05857527
Title: Extending taVNS Paired With Infant CIMT Into a Home-Based Setting: Technology Development Requisite for a Randomized Trial
Brief Title: Extending taVNS Paired With Infant CIMT Into a Home-Based Setting
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00123579
Record Dates: First submitted 2023-02-23; First posted 2023-05-12 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Laboratories; Home Care Services

STUDY DESIGN:
Intervention Model Description: For this study we are making modifications to the taVNS stimulation (Soterix unit) system. These modifications include using Electromyography (EMG) muscle sensors to trigger stimulation instead of a manual button. We are also transitioning the manual stimulation option to Bluetooth to improve ease of use in the clinic with infants. The taVNS stimulation will be paired with constraint induced movement therapy (CIMT) an established rehabilitation intervention. The Soterix taVNS unit is FDA registered and is a custom version of an FDA cleared device. The first 2 participants will complete phase 1 of the study. In this phase we will make adjustments to the EMG system and physical set up with the goal of having the EMG sensors trigger taVNS stimulation with 75% of total time for active arma and trunk movements during CIMT. In phase 2 we will use the EMG triggered taVNS setup to deliver CIMT in home.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EMG triggering feasibility (Experimental): We will trial use of a new taVNS unit that uses automated EMG sensors to trigger stimulation and an optional Bluetooth manual trigger. This experimental device will be used to during CIMT rehabilitation treatment to pair stimulation with active movement.
  Interventions: Combination Product: Custom EMG triggered Soterix taVNS stimulation with CIMT therapy in lab
- taVNS and EMG feasibility at home (Experimental): For the 2nd phase of the study we will trial using the EMG triggered system to deliver taVNS and CIMT in the home setting.
  Interventions: Combination Product: Custom EMG triggered Soterix taVNS stimulation with CIMT therapy in home

INTERVENTIONS:
Combination Product: Custom EMG triggered Soterix taVNS stimulation with CIMT therapy in lab — Participants will receive taVNS stimulation paired with 40 hours of constraint-induced movement therapy. The new device will automatically trigger stimulation using EMG muscle sensors worn during the therapy session. Phase 1 will occur in the lab, and ongoing notifications will be made to the EMG system to test feasibility of automatic stimulation
  Arms: EMG triggering feasibility
Combination Product: Custom EMG triggered Soterix taVNS stimulation with CIMT therapy in home — Participants will receive taVNS stimulation paired with 40 hours of constraint-induced movement therapy. The new device will automatically trigger stimulation using EMG muscle sensors worn during the therapy session. Phase 2 will occur in the home and will assess the quality of the CIMT therapy provided with the automated EMG system.
  Arms: taVNS and EMG feasibility at home

SUMMARY:
Newborns who are born premature or suffer brain injury at birth are at risk for motor problems that may cause weakness in reaching and grasping on one side of the body. In older children, therapists may use a hand mitt and restraint for the stronger arm, to encourage use of the weaker side, called constraint-induced movement therapy (CIMT). Even with the high intensity therapy of CIMT, it typically takes between 40-120 hours total treatment time for most children to improve their motor skills. A non-invasive form of nerve stimulation, transcutaneous auricular vagus nerve stimulation (taVNS), stimulates a nerve by the ear that enhances learning motor skills. taVNS stimulation will be triggered by EMG sensors which detect muscle activity. The purpose of this study is to evaluate the safety and effectiveness of taVNS to improve motor skills when paired with CIMT in infants with one-sided weakness at 6-18 months of age.

DETAILED DESCRIPTION:
Preterm birth and complications in term births can result in increased risk for intraventricular hemorrhage, global hypoxia-ischemia (HIE), arterial stoke, and neuroinflammation with white matter injury in newborns. Centeral Nervous System (CNS) injuries then may manifest as early developmental delays and motor weakness in the first 12 months, that presage hemiplegic cerebral palsy (CP).

Early targeted therapy interventions for high-risk infants aim to improve neurological outcomes by taking advantage of critical windows for neuroplasticity. Intensive interventions, such as constraint-induced movement therapy (CIMT), are designed to ameliorate early motor predecessors of CP in at-risk infants. This intervention must be provided at a minimally effective dosage of 40 hours, and 60-120 hours for optimal outcomes, and are typically provided in a condensed time period, over 4 to 6 weeks with intensive task-practice for 3-6 hours a day. Delivering CIMT within the context a typical family day is a challenge. Interventional strategies that reduce the time requirement while offering the same or better outcomes would benefit families and facilitate treatment delivery.

Few studies have used neuromodulation combined with intensive motor therapies, such as CIMT, to enhance neuroplasticity and improve functional outcomes in children. Transcranial direct current stimulation has been used safely in older children with CP during bimanual learning therapy. Our group is the first to use non-invasive transcutaneous auricular vagus nerve stimulation (taVNS) paired with a motor task of bottle-feeding in infants with feeding failure. taVNS paired with motor feeding activity was safe and over 50% infants determined to need a gastrostomy tube (G-tube) attained full oral feeds (mean time to full oral feeds 15 days with once daily, and 7.8 days with twice daily treatment). This study will use EMG sensing of muscle activity to trigger the taVNS system. Use of EMG sensors is hypothesized to improve pairing of stimulation with motor activity while also decreasing the treatment burden for the therapist.

ELIGIBILITY:
Inclusion Criteria:

* Five 6-18-month-old infants
* Hemiplegia/motor asymmetry qualifying for Constraint Induced Movement Therapy
* Gross Motor Function Classification System (GMFCS) level I-IV
* Ability to maintain a sitting position for 5 minutes with moderate assistance

Exclusion Criteria:

* GMFCS level V
* Severe motor impairment/ quadriplegic involvement
* Uncorrected blindness or deafness
* Cardiomyopathy

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred through flyers in the local hospital and clinics. Flyers were provided to high-risk infant follow-up clinics to be distributed to eligible parents.
Pre-assignment Details: All participants received 40 hours of CIMT paired with taVNS. The first 2 participants received treatment in the lab so the engineer could address sensor calibration and settings to automate EMG triggering. The remaining participants received the same 40 hours of CIMT paired with taVNS in the home setting with the goal to test feasibility of translation of the new EMG triggered taVNS into standard home therapy settings. Participants were told if they would be in home or lab before consent.
Groups:
- Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Lab: Participants will receive taVNS stimulation paired with 40 hours of constraint-induced movement therapy. The new device will automatically trigger stimulation using EMG muscle sensors worn during the therapy session. Phase 1 will occur in the lab, and ongoing notifications will be made to the EMG system to test the feasibility of automatic stimulation
Period: Overall Study
Arm/Group | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Lab | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Home
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Lab | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Home | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: months] | 18.5 [18 to 19] | 22.5 [22 to 23] | 20.5 [18 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
Gross Motor Functional Measure (GMFM) function at baseline [Mean (Full Range); unit: Gross Motor Functional Measure 66 score] — Gross Motor Functional Measure The GMFM consists of 5 domains: a)Lying & Rolling, b)Sitting, c)Crawling & Kneeling, d) Standing, and e) Walking, Running & Jumping. Each item in the test uses a 4-point scale: 0=does not initiate; 1=initiates but completes less than 10%; 2=partially completes (10% to less than 100%); and 3=fully completes the task.
  Item scores are summed to calculate raw and percent scores for each of the five domains. Domain percent scores are averaged to obtain an overall total score. Higher scores represent higher levels of function. The total score range is 0 to 100%.
  Gross Motor Functional Measure 66 score | 36 [27 to 45] | 31.5 [23 to 40] | 33.75 [23 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Device Feasibility
Description: Feasibility is measured as percent of total treatment time Electromyography (EMG) can successfully trigger stimulation during a Constraint induced movement therapy (CIMT) rehabilitation session.
Time Frame: end of 4 week treatment intervention (40 hours of CIMT)
Measure: Mean (Full Range); unit: percent time EMG taVNS stimulation
Arm/Group | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Lab
Number analyzed (Participants) | 2
percent time EMG taVNS stimulation | 33.33 [3 to 77]

2. Secondary Outcome: Fidelity of Implementation Measure (FIRM)
Description: Fidelity Rating of Quality of Constraint Induced Movement Therapy Delivery while using the experimental EMG triggered Soterix taVNS stimulator.
  Fidelity of Implementation Measure (FIRM) which describes how consistently therapists exhibit behaviors consistent with CIMT principles and operant conditioning techniques and are rated on a scale of 1-4. A 4 being consistently demonstrating with less than 1 exception, and 1 being rarely or not at all. A score of 3 indicates acceptable to high fidelity.
Time Frame: end of 4 week treatment intervention (40 hours of CIMT)
Population: Even though we met the threshold to move to trialing the EMG triggered taVNS in home we faced technical issues with the EMG triggering interface. We completed the full 40 hours of CIMT therapy but could not use EMG triggered taVNS stimulation. Therefore, we were not able to rate the fidelity of the CIMT treatment with TMG triggered taVNS because the EMG system did not function properly. Our 2nd participant withdrew and therefore, we were again not able to rate the fidelity of implementation.
Arm/Group | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Home
Number analyzed (Participants) | 0

3. Secondary Outcome: Quality of Upper Extremity Skills Test (QUEST)
Description: Quality of Upper Extremity Skills Test The QUEST is a criterion-referenced measure designed to evaluate the quality of upper extremity function in young children with spasticity. We calculated scores from 2 domains:1) Dissociated movement and2) Grasp Item scores are summed; formulas are used to calculate percentages for each domain. Domain percentages are summed and divided by number of domains (2 for our study) to obtain total score. Minimum score = 0; Maximum score = 100 The total QUEST score was calculated by summing scores for each sub-domain tested divided by the total number of sub-domains tested. The total scores on the QUEST range from 0 to 100. Higher scores represent better quality of movement.
Time Frame: Change in functional motor outcome completed pre and post 40 hours of treatment
Population: We completed analysis on the 3 participants who received 40 hours of CIMT therapy paired with taVNS. The 2nd participant in the home group withdrew and did not complete the 40 hours of therapy so change in function was not assessed.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Lab | Custom EMG Triggered Soterix taVNS Stimulation With CIMT Therapy in Home
Number analyzed (Participants) | 2 | 1
score on a scale | 14.8 [8.01 to 21.59] | 24.89 [24.89 to 24.89]

ADVERSE EVENTS:
Time Frame: Study staff were in daily contact with participants throughout treatment. After the 4 week interventions, we followed up at 3 months up to 4 months post for final assessments.
Groups:
- Soterix taVNS Stimulation Using EMG Sensors: We will trial use of a new taVNS unit that uses automated EMG sensors to trigger stimulation and an optional Bluetooth manual trigger. This experimental device will be used to during CIMT rehabilitation treatment to pair stimulation with active movement.
  Custom EMG triggered Soterix taVNS stimulation with CIMT therapy: Participants will receive taVNS stimulation paired with 40 hours of constraint-induced movement therapy. The new device will automatically trigger stimulation using EMG muscle sensors worn during the therapy session.
Arm/Group | Soterix taVNS Stimulation Using EMG Sensors
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The purpose of this trial was to test the feasibility of using EMG to trigger taVNS stimulation. The EMG sensors did not stay in place well for some infants. Additionally, there was a large amount of time and effort required for individual calibration. We met the goal threshold of phase 1 for our EMG sensor to trigger taVNS stimulation. However, the automatic triggering did not continue to work well for subsequent participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT05857527/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT05857527/ICF_000.pdf